CLINICAL TRIAL: NCT00003786
Title: A Phase II Trial of MGI-114 (NSC# 683863) Administered as a 5-Minute Infusion Daily for Five Days Every 4 Weeks in Patients With Previously Untreated Advanced Colorectal Cancer
Brief Title: Irofulven in Treating Patients With Metastatic or Recurrent Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: NO participants
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9635; UCCRC-9635; NCI-T98-0008
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — irofulven

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): MGI-114 (11mg/m2/day x 5 days every 28 days)
  Interventions: Drug: irofulven

INTERVENTIONS:
Drug: irofulven

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irofulven in treating patients with metastatic or recurrent colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate of patients with metastatic or locally recurrent adenocarcinoma of the colon or rectum treated with 6-hydroxymethylacylfulvene (MGI-114). II. Determine the toxicity of this treatment regimen in this patient population. III. Study pharmacokinetics of MGI-114 in these patients. IV. Determine the relationship between pharmacokinetics of MGI-114 and clinical outcomes including toxicity and response to therapy in these patients.

OUTLINE: This is an open label, multicenter study. Patients receive 6-hyroxymethylacylfulvene (MGI-114) IV over 5 minutes daily for 5 days. Courses are repeated every 4 weeks. Treatment continues for a minimum of 2 courses in the absence of unacceptable toxic effects or disease progression. Patients are followed until death.

PROJECTED ACCRUAL: A total of 14-35 patients will be accrued for this study within 6-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic or locally recurrent adenocarcinoma of the colon or rectum Bidimensionally measurable disease Lesions seen on colonoscopic examination or barium studies, bone metastases, CNS lesions, CEA levels and ascites are not considered measurable No CNS disease only CNS metastases with other sites of measurable disease allowed provided appropriate therapy for CNS metastases has been administered and patient is neurologically stable and does not require intravenous steroid or anticonvulsant therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 OR Zubrod 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3,500/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 (no platelet transfusion within 7 days) Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No significant uncontrolled medical or psychiatric illness No serious active infection No other active malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix unless adequately treated and less than 30% risk of relapse

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent prophylactic use of growth factors except for documented febrile neutropenia or sepsis Chemotherapy: At least 12 months since prior fluorouracil based adjuvant or neoadjuvant chemotherapy No more than 1 prior regimen No prior chemotherapy for advanced metastatic colorectal cancer No other concurrent chemotherapy No concurrent investigational antineoplastic drugs Endocrine therapy: See Disease Characteristics Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No prior radiotherapy to the only site of measurable disease No concurrent radiotherapy Surgery: Not specified Other: See Disease Characteristics At least 30 days since prior investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-04; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Clinical Response Rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L. Kindler, MD, Study Chair — University of Chicago
Locations (9):
- United States (9):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Illinois Oncology Research Association, Peoria, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana
  - James Graham Brown Cancer Center, Louisville, Kentucky